CLINICAL TRIAL: NCT05995548
Title: Mechanisms Involved in the Developement of Sports Addiction Among Military Personnel
Acronym: DEEP_SPORT
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PPRC09; 2023-A00013-42 (Other: IDRCB)
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Addiction
Keywords: Sports addiction; Military; Comprehension model
MeSH Terms: conditions — Behavior, Addictive | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — The interview will take place face-to-face. It will take place in a quiet room, with the door and windows closed. Only the participant and the investigator will be present. It will be recorded using a dedicated to this research. At the end of the interview, so as not to influence the participant's discourse, the participant will be asked to fill in the self-questionnaire 'EAI' (Exercise Addiction Inventory), which will confirm or refute the diagnosis, thus exploring a possible discrepancy between the participant's feelings and the diagnosis.

SUMMARY:
Sport addiction (or exercise addiction) has been recognized as a pathology by the World Health Organization since 2011. However, it is still relatively under-researched. It is one of the so-called behavioral addictions and has long-term negative consequences for physical, psychological and social health, such as : isolation ; frequent injuries; co-addiction with or as a result of sports'.

The study is aimed in particular at military physicians and will target a population where sport is an integral part of the job and where sporting performance is valued: military personnel.

The aim of this study is to explain and try to understand this pathology through the experiences of those who suffer from it. Therefore, investigators have chosen to conduct a qualitative study inspired by the embedded theory. Semi-structured individual interviews will be conducted using an interview guide. This guide, consisting of 5 or 6 open-ended questions, will help to set the general direction of the interview without preventing the participant from deviating. The interview guide may evolve as the interviews progress, enriched by any new ideas or themes that emerge.

ELIGIBILITY:
Inclusion Criteria:

* Serving or reservist military personnel
* Perceive themselves as "addicted to sport" and say so

Exclusion Criteria:

* Minor
* Incapable major
* Patient unaware of diagnosis
* Pregnant woman
* Legionnaire not rectified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of sport addicts military subjects.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Explanatory model | Through study completion (30 months)
  The primary outcome is to propose an explanatory model for sport addiction in the military personnel.

CONTACTS AND LOCATIONS:
Locations (1):
- CMA09, Hyères, France

IPD SHARING:
Plan to Share IPD: No